CLINICAL TRIAL: NCT00006068
Title: Does Islet Transplantation Eliminate Hypoglycemia?
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: National Center for Research Resources (NCRR) (NIH)
Allocation: Non-Randomized | Masking: Single | Purpose: Treatment
Other Study IDs: NCRR-M01RR00036-0746; M01RR000036 (NIH)
Record Dates: First submitted 2000-07-18; First posted 2000-07-19 (Estimated); Last update posted 2005-06-24 (Estimated); Status verified 2001-11

CONDITIONS: Diabetes Mellitus
MeSH Terms: conditions — Diabetes Mellitus | interventions — Islets of Langerhans Transplantation

INTERVENTIONS:
Procedure: Pancreatic Islet Transplantation

SUMMARY:
Low blood sugar (hypoglycemia) is a recurrent problem for many people with diabetes. Successful transplantation of clusters (islets) of normal cells, that include those which produce the sugar-lowering hormone insulin, from the pancreas of a person who did not have diabetes into a person with diabetes should eliminate high blood sugar levels. We wish to determine if it will also eliminate low blood sugar. To do so we will give insulin to lower the blood sugar, measure the levels of the hormones that normally raise blood sugar levels (e.g., glucagon and epinephrine) and then stop the insulin and see if blood sugar levels return to normal. Because we anticipate that the transplanted islets will produce insulin, but not glucagon, this study may also tell us if regulated insulin production alone can prevent hypoglycemia in humans.

ELIGIBILITY:
Inclusion Criteria:

* Clinically stable, insulin dependent islet transplant recipients and matched nondiabetic healthy controls

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult